CLINICAL TRIAL: NCT01448525
Title: Study Assessing Patient Satisfaction With LATISSE® for Increasing Eyelash Prominence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GMA-LTS-11-002
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-04

CONDITIONS: Hypotrichosis
MeSH Terms: conditions — Hypotrichosis | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bimatoprost ophthalmic solution 0.03% (Active Comparator): One drop of bimatoprost ophthalmic solution 0.03% applied to the upper eyelid margin of both eyes once daily in the evenings for 16 weeks.
  Interventions: Drug: bimatoprost ophthalmic solution 0.03%
- bimatoprost vehicle solution (Placebo Comparator): One drop of bimatoprost vehicle solution applied to the upper eyelid margin of both eyes once daily in the evenings for 16 weeks.
  Interventions: Drug: bimatoprost vehicle solution

INTERVENTIONS:
Drug: bimatoprost ophthalmic solution 0.03% — One drop of bimatoprost ophthalmic solution 0.03% applied to the upper eyelid margin of both eyes once daily in the evenings for 16 weeks.
  Other Names: LATISSE®
  Arms: bimatoprost ophthalmic solution 0.03%
Drug: bimatoprost vehicle solution — One drop of bimatoprost vehicle solution applied to the upper eyelid margin of both eyes once daily in the evenings for 16 weeks.
  Arms: bimatoprost vehicle solution

SUMMARY:
The purpose of this study is to determine patient satisfaction with LATISSE® treatment for increasing eyelash prominence.

ELIGIBILITY:
Inclusion Criteria:

* Have inadequate eyelashes
* Never used prescription eyelash growth products

Exclusion Criteria:

* No visible eyelashes
* Permanent eyeliner or eyelash implants
* Semi-permanent eyelash tint, dye, or extensions within 3 months
* Over-the-counter eyelash growth products within 6 months
* Any disease, infection or abnormality of the eye or area around the eye
* Eye surgery within 3 months, or the anticipated need for eye surgery during the study
* Unable or unwilling to keep contact lenses out during drug application and for 30 minutes after application

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Coral Gables, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Bimatoprost Vehicle Solution
Started | 44 | 44
Completed | 43 | 42
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Bimatoprost Vehicle Solution | Total
Number analyzed (Participants) | 44 | 44 | 88
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (12.6) | 50.2 (10.5) | 49.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Satisfied or Very Satisfied With Their Eyelashes Overall
Description: Participants rated their overall eyelash satisfaction by answering Eyelash Satisfaction Questionnaire (ESQ-9) question #3: "Overall, how satisfied are you with your eyelashes?" using a 5-point scale: -2=very unsatisfied (worst), -1=unsatisfied, 0=neutral, 1=satisfied or 2=very satisfied (best). The percentage of participants who rated their satisfaction as 1=satisfied or 2=very satisfied at Week 16 is reported.
Time Frame: Week 16
Population: Intent to treat population included all randomized participants who had at least 1 post-baseline efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 43 | 42
Percentage of participants | 67.4 | 7.1

2. Secondary Outcome: Percentage of Participants With at Least a 1-Grade Increase in the Global Eyelash Assessment (GEA) Score
Description: The investigator evaluated the patient's overall eyelash prominence using the 4-point GEA scale: 1=minimal (worst), 2=moderate, 3=marked or 4=very marked (best). An at least a 1-grade increase in GEA score indicated improvement.
Time Frame: Baseline, Week 16
Population: Intent to treat population included all randomized participants who had at least 1 post-baseline efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 43 | 42
Percentage of participants | 72.1 (0.37) | 19.0 (0.43)

ADVERSE EVENTS:
Description: Treatment-emergent adverse events are presented.
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Bimatoprost Vehicle Solution
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 1/44 | 3/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Ophthalmic Solution 0.03% (N=44) | Bimatoprost Vehicle Solution (N=44)
Nasopharyngitis (Infections and infestations) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.